CLINICAL TRIAL: NCT03574272
Title: Demonstration and Multi-center Verification of the Patient Transfer Monitoring System in Hospital Using Mobile IoT Technology
Brief Title: Patient Transfer Monitoring System in Hospital Using Mobile IoT Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Korea Health Industry Development Institute (Other Government)
Responsible Party: Principal Investigator, Chang-Min Choi, associate professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C2018-00554
Record Dates: First submitted 2018-05-27; First posted 2018-06-29 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Patient Monitoring
Keywords: mobile IoT technology; Patient Transfer Monitoring System

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient Transfer Monitoring System (Experimental)
  Interventions: Other: Patient Transfer Monitoring System

INTERVENTIONS:
Other: Patient Transfer Monitoring System — The subjects will be provided with portable oximeter and smart-phone which application for monitoring is installed, and the transmitted data will be monitored in real time via monitoring equipment in the (Patient-hospitalized) ward.

SUMMARY:
This trial is multi-center prospective study to develop Patient Transfer Monitoring system using mobile lot network and the Risk Factor Detection System and apply to real In-Hospital Patients and verify the efficacy.

DETAILED DESCRIPTION:
Hospitalized patients who need transfer for a diagnostic examination or rehabilitation therapy during hospitalization, and have a risk of hypoxemia during transfer will be enrolled in this trial. The subjects will be provided with a portable oximeter and a smart-phone which application for monitoring is installed, and oxygen saturation and pulse rate will be checked in real time during transfer. The collected data will be transferred to cloud system via Iot network, and the transmitted data will be monitored in real time via monitoring equipment in the (Patient-hospitalized) ward. If there is a risk, the alarm system is activated so that the medical team is able to check risk factor and manage it immediately.

All the risk factors and severity will be collected during transfer, also these are checked whether the monitoring system and the data transmission system work properly or not, the time from detecting risk factor to medical response, the composition of medical staffs who responding to alarmed risk factors and improvement of the subjects.

Pilot study will be conducted with 20 subjects in Asan medical center. In pilot study, monitoring machines (HR, SpO2 monitor) commonly used in wards or hospitals will be used to verify the stability of oximeter used in this study and the developed risk detection system.

ELIGIBILITY:
Inclusion Criteria:

* A hospitalized patients in pulmonology department or rehabilitation hospital who have a risk of decreasing oxygen saturation
* A patients who require transfer in the hospital for a diagnostic examination or rehabilitation therapy during hospitalization
* Patients who need oxygen saturation monitoring according to the investigator's judgment
* Patients who voluntarily agree to study participation and provide written informed consent form

Exclusion Criteria:

* Patients who don't agree with the study procedure or are uncooperative
* Repeated monitoring of the same patient who already registered in the tiral

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2018-05-16 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2018-12-28 (Actual)

PRIMARY OUTCOMES:
frequency of risk factors which are detected during transfer | from the beginning to immediately after the end of the patient transfer
severity of risk factors which are detected during transfer | from the beginning to immediately after the end of the patient transfer
  The severity is assessed as mild(risk factor was resolved without medical staff), moderate(resolved by medical staffs, but returned to the ward), and severe(not resolved by medical staffs, needs other method such as CPCR call, invasive intervention).
reason of decreased oxygen saturation | from the beginning to immediately after the end of the patient transfer
duration of decreased oxygen saturation | from the beginning to immediately after the end of the patient transfer
change from baseline in Oxygen saturation | from the beginning to immediately after the end of the patient transfer
the time from detecting risk factor to medical response | from the beginning to immediately after the end of the patient transfer
Death | from admission to discharge, up to 8 months
admission to intensive care units | from admission to discharge, up to 8 months
Adverse events related to the study | from the beginning to immediately after the end of the patient transfer
medical staffs who managed the alarmed event during transfer | from the beginning to immediately after the end of the patient transfer

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Min Choi, MD, Ph. D, Principal Investigator — Asan Medical Center
Locations (5):
- South Korea (5):
  - Kangwon National Univeristy Hospital, Chuncheon, Gangwon-do
  - DAVINCI hospital, Daejeon
  - KyungHee University Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Wonju Severance Christian Hospital, Wŏnju

IPD SHARING:
Plan to Share IPD: Undecided